CLINICAL TRIAL: NCT06082128
Title: Improving the Wellbeing of People With Advanced Cancer and Their Family Carers: An Effectiveness Implementation Trial of an Australian Dyadic Digital Health Intervention (FOCUSau)
Brief Title: FOCUSau: A Dyadic Digital Health Intervention to Improve the Wellbeing of People With Advanced Cancer and Their Carers
Acronym: FOCUSau
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Melbourne (Other)
Collaborators: St Vincent's Hospital Melbourne (Other); University of Technology, Sydney (Other); National Health and Medical Research Council, Australia (Other); University of Sydney (Other); Peter MacCallum Cancer Centre, Australia (Other); Vrije Universiteit Brussel (Other); Flinders University (Other); Queensland University of Technology (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 84479; APP2006170 (Other Grant/Funding Number: National Health and Medical Research Council (NHMRC))
Record Dates: First submitted 2023-09-20; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Advanced Cancer
Keywords: Palliative care; End-of-life decision making; Supportive care; Psychoeducational intervention; Dyadic; Family caregiver; Quality of life

STUDY DESIGN:
Masking Description: Due to the nature of the intervention the dyads cannot be blinded to allocation. The research nurse/officers involved in the consenting process will not be blinded as they will facilitate the second videoconference to inform the dyads about their allocated group (intervention or control). As data collection will occur electronically (via the FOCUSau platform) the research team will be blinded to which trial group the dyads were randomised to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Dyads in the control group will receive usual care only. Usual advanced cancer care is known to be heterogeneous. It is expected usual care to include care from specialists, doctors, nurses or other health care professionals that patients usually engage with.
- FOCUSau (Experimental): Dyads in the FOCUSau arm will receive the web-based FOCUSau program in addition to usual care.
  Interventions: Behavioral: FOCUSau

INTERVENTIONS:
Behavioral: FOCUSau — FOCUSau is a self-administered web-based intervention and completed autonomously via the internet by the dyad. Delivery encompasses the completion of four prescribed consecutive FOCUSau sessions (with three weeks between each session) over a period of 12 weeks.
  The sessions are completed simultaneously by the patient and family carer, together at a computer. The intervention sessions can be completed at any time within the 12-week timeframe. Participants receive tailored individual and dyadic messages according to the information provided at study enrollment and their responses to questions within the sessions. Dyads are also provided with an online personal workbook containing the results of interactive exercises completed during the internet sessions. Any information sheets that the dyad indicated as 'of interest to them' during the internet sessions are included as a hyperlink in their personal workbook which also contains evidence-based local advanced cancer related resources.
  Other Names: Family involvement(F),Supporting outlook and meaning(O),Increasing Coping Effectiveness(C),Reducing Uncertainty(U),Symptom Management(S); FOCUSau (web-based intervention)
  Arms: FOCUSau

SUMMARY:
FOCUS is a dyadic, psychoeducational intervention developed in the USA, shown to improve the wellbeing and quality of life (QoL) of patients with advanced cancer and their primary family carers. The intervention consists of five core components underpinning the FOCUS acronym:

(F) supporting Family involvement, (O) supporting Outlook and meaning, (C) increasing Coping effectiveness, (U) reducing Uncertainty, and (S) Symptom management. Originally a nurse-delivered in-person intervention, FOCUS has been translated into a self-administered web-based intervention as part of an European study.

The overall aim of this project is to determine the effectiveness and sustainability of a digital health intervention (FOCUSau) aimed at improving the wellbeing and self-efficacy of patients with advanced cancer and their primary support person/carer.

A primary support person/carer is an unpaid individual identified by the person with advanced cancer (not necessarily a partner or family member) who is providing them with physical, social or emotional support. Hereafter referred to as a "carer". The term "dyad" refers to the patient and primary support person/carer.

The project objectives are:

1. adapt FOCUS to the Australian context and develop FOCUSau;
2. examine the effectiveness of FOCUSau in improving the wellbeing (primary outcomes: QoL and self-efficacy) of patients with advanced cancer and their primary family carer;
3. compare the type and costs of health service use by participants in the intervention and control group; and
4. assess the acceptability, feasibility and scalability of FOCUSau in order to inform sustainable implementation of the intervention within the Australian health care system.

A pragmatic phase III hybrid effectiveness-implementation trial with an integrated research design that includes digital health evaluation will be used in patients with advanced cancer and their primary support person/carer.

Data will be collected three times from patient-carer dyads:

1. at baseline (T0) after which the dyad will immediately be randomised to one of the study arms,
2. first follow-up at 12 weeks after baseline (T1) and,
3. second follow-up at 24 weeks after baseline (T2).

DETAILED DESCRIPTION:
STUDY SETTING:

The patient-carer dyads will be recruited via two methods: (1) referral from hospitals or (2) self-referral. For method one, approximately six hospitals and/or cancer centres (metropolitan and regional) across Australia will be selected. For the self-referral recruitment method, patients who have been made aware of the project (but have not been officially screened by a clinician) may self-refer via a webform on the project website. These patients will be made aware via consumer/carer/cancer advocacy groups, or social media advertisement.

SAMPLE SIZE:

A pre-determined strict fixed sequence (FS) procedure defines prospectively hierarchical ordering of the primary endpoints; emotional wellbeing (1) and self-efficacy (2). Testing of null hypotheses proceeds according to their hierarchical order; that is, hypothesis 1 (H(1)0) is tested first at a significance level of 5%, and if H(1)0 is rejected then hypothesis 2 (H(2)0) is tested at the same significance level, otherwise H(2)0 is not tested at all. The strict FS approach has the highest power for testing the first hypothesis (outcome: emotional wellbeing) compared to the other methods, as it does not save any portion of alpha for testing later hypothesis. The reference mean value from The European Organization for Research and Treatment of Cancer (EORTC) for all cancer patients, stage III-IV is 71.5 (SD: 23.8). To maintain rigorous control over Type I errors due to multiple comparisons, the alpha level is set at 0.025 instead of the more common 0.05. This adjustment accounts for the multiple comparisons required in the study, including comparisons between a control group and two participant groups (patients and carers). Statistical power is set at 0.80. The expected difference between the control group and the intervention arm in the primary outcomes is 0.375 SD at T1 (12 weeks). With these parameters n=173 dyads are needed in each arm (i.e. 346 dyads in total). Anticipating a maximum 80% retention rate at T1 (USA FOCUS retention was 86%) approximately 433 dyads will need to be recruited. An enrolment rate of 55% of those eligible was achieved in prior digital health FOCUS study from 2014, however it is anticipated this will be higher for FOCUSau (estimating 70%) given the internet is much more widely available now and the digital recruitment approach; meaning that approximately 618 dyads who meet eligibility criteria will need to be identified. Evidence also suggests that recruitment rates can increase when a digital health intervention is offered.

DATA ANALYSIS:

The effectiveness of FOCUSau will be compared with the standard care (control group) for each participant population (patients/carers) using significance level of alpha=0.025. The hypotheses will be tested using a mixed model (per participant population) with the T1 measurement values for emotional wellbeing and self-efficacy as primary outcomes. These mixed models will be implemented using International Business Machines Corporation (IBM) Statistical Package for the Social Sciences (SPSS) for Windows Version 27.0 and R with recruitment centre treated as a random effect and randomisation group as predictor variables. As per the fixed sequence (FS) procedure, the null hypotheses of the second primary endpoint (self-efficacy) will only be tested if a significant result is found for the first primary endpoint (emotional wellbeing). Additionally, other factors identified in the literature will be incorporated as potentially predictive by including them as covariates in the mixed models. Analyses on both 'intention-to-treat' and per-protocol principles will be performed. To interpret the magnitude of the effects for the different outcomes, effect sizes will be estimated (Cohen's d).

The data analysis will encompass all primary and secondary outcomes. Primary endpoints, including emotional wellbeing and self-efficacy measured at T1, will be analysed first. Following that, secondary endpoints, comprising outcomes measured at T1 that are not primary endpoints, as well as all outcomes measured at T2 (occurring 24 weeks from T0), will be assessed. This approach allows for a comprehensive evaluation, including the examination of longer-term effects.

The robustness and validity of the results will be explored using sensitivity analyses by varying the parameter inputs (including sensitivity to the use of values for missing observations). The analysis will be conducted for the within trial period; the potential to extrapolate results over the longer-term will be assessed based on the proportion of patients alive at the end of follow-up.

The cost-effectiveness analysis will be reported as the mean costs of care per dyad in each arm of the study. Costs applied to health care service use will be as per Australian standard fees (e.g., via the Medicare Benefits Schedule). If a difference in outcomes is observed, as hypothesised, the incremental cost effectiveness of FOCUSau compared with control will be estimated in terms of the: (1) cost per additional patient with a meaningful improvement in emotional wellbeing (as assessed using the EORTC QLQ-C30 emotional wellbeing scale); and separately, (2) cost per additional carer with a meaningful change in self-efficacy (as assessed using the The Lewis´ Cancer self-efficacy scale). The base case analysis of cost-effectiveness will be conducted from a health care system perspective. Subsequent sensitivity analyses will modify the assessment of costs to adopt a societal perspective to capture the impact of informal care costs, as well as testing the robustness of the analysis results to variations in other parameter inputs.

Missing data for costs and outcomes will be described and summarised. Where missing data can be regarded as missing at random, likelihood (interpolation) methods will be used for analysis of those data as appropriate.

ELIGIBILITY:
Patient Inclusion Criteria:

* Diagnosis of advanced cancer
* Over 18 years of age
* Able to comprehend written or spoken English
* No visual, hearing, and/or cognitive impairment that would preclude participation
* Able to commit to research participation requirements (including data collection and completion of the FOCUSau intervention if randomised to that group)
* Able to access the internet (on desktop computer, laptop computer or tablet device)
* Able to identify a primary support person/carer, who is an unpaid individual (not necessarily a partner or family member) who is providing physical, social or emotional support.

Patient Exclusion Criteria:

- Involvement in an advanced cancer non-drug trial that focuses on improving QoL

Family carer Inclusion Criteria:

* Identified by the patient as their primary support person who is related to them biologically, legally or emotionally, and is willing to accept this support role
* Aged over 18 years
* No visual, hearing, and/or cognitive impairment that would preclude participation
* Able to commit to research participation requirements
* Able to access the internet

Dyad Inclusion Criteria:

- Capacity to effectively utilise the internet (as determined through a short practical online exercise as part of the screening and consent process).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in emotional wellbeing | T0 (baseline), T1 (12 weeks) and T2 (24 weeks)
  For patients and for carers: The European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) 10 emotional function items
Change in self-efficacy | T0 (baseline), T1 (12 weeks) and T2 (24 weeks)
  For patients and for carers: The Lewis´ Cancer self-efficacy scale

SECONDARY OUTCOMES:
Change in patient quality of life | T0 (baseline), T1 (12 weeks) and T2 (24 weeks)
  For patients: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 15 Palliative Care (EORTC QLQ-C15-PAL)
Change in carer quality of life | T0 (baseline), T1 (12 weeks) and T2 (24 weeks)
  For carers: The Caregiver Quality of Life Index-Cancer (CQOLC)
Change in patient social wellbeing | T0 (baseline), T1 (12 weeks) and T2 (24 weeks)
  For patients: social wellbeing scale from Functional Assessment of Cancer Therapy - General (FACT-G)
Change in patient social functioning | T0 (baseline), T1 (12 weeks) and T2 (24 weeks)
  Two social functioning items from The European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30
Change in patient overall health | T0 (baseline), T1 (12 weeks) and T2 (24 weeks)
  Two items about overall health from The European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30
Change in appraisal of illness | T0 (baseline), T1 (12 weeks) and T2 (24 weeks)
  For patients and for carers: Benefits of Illness Scale
Change in coping | T0 (baseline), T1 (12 weeks) and T2 (24 weeks)
  For patients and for carers: A shortened version of Brief Cope
Change in ways of giving support | T0 (baseline) T1 (12 weeks) T2 (24 weeks)
  For patients and for caregivers: The five items 'Active engagement scale' from the ´Ways of giving support questionnaire´
Change in dyadic coping | T0 (baseline) T1 (12 weeks) T2 (24 weeks)
  For patients and for caregivers: Three scales from the 'Dyadic Coping Inventory': 'Stress communication by oneself', 'Stress communication by partner' and 'Evaluation of dyadic coping'
Patient level of functioning | T0 (baseline), T1 (12 weeks) and T2 (24 weeks)
  Modified version of Eastern Cooperative Oncology Group (ECOG) Performance Status Assessment
Change in utilisation of healthcare and associated services | T0 (baseline), T1 (12 weeks) and T2 (24 weeks)
  For patients and for caregivers: Client Service Receipt Inventory (CSRI)
Change in quality-adjusted life years | T0 (baseline), T1 (12 weeks) and T2 (24 weeks)
  For patients and for caregivers: EuroQoL EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hudson, PhD, Principal Investigator — The University of Melbourne and St Vincents Hospital Melbourne
Locations (5):
- Australia (5):
  - Calvary Healthcare Kogarah, Kogarah, New South Wales
  - Mater Health Service, Kangaroo Point, Queensland
  - Northern Adelaide Palliative Service, Modbury, South Australia
  - Barwoon Health Mckellar Centre, Geelong, Victoria
  - St Vincents Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
Results will be published in peer-reviewed, international journals. Local and International conference presentations are anticipated. Opportunities for sharing the study results via media will be sought (e.g., social media platforms such as Twitter).
  An option will be provided to participants to receive a plain language summary of the study results. We will use this plain language summary to provide the study results to relevant consumer networks including the Victorian Comprehensive Cancer Centre and Cancer Voices Australia.

REFERENCES:
- [Derived] Hudson P, Francis J, Cohen J, Kapp S, De Abreu Lourenco R, Beatty L, Gray K, Jefford M, Juraskova I, Northouse L, de Vleminck A, Chang S, Yates P, Athan S, Baptista S, Klaic M, Philip J. Improving the Well-Being of People With Advanced Cancer and Their Family Caregivers: Protocol for an Effectiveness-Implementation Trial of a Dyadic Digital Health Intervention (FOCUSau). JMIR Res Protoc. 2024 Aug 13;13:e55252. doi: 10.2196/55252. PMID 39137414